CLINICAL TRIAL: NCT02948088
Title: A Disease Registry for Patients With Tenosynovial Giant Cell Tumors (TGCT), Also Known as Pigmented Villonodular Synovitis (PVNS) and Giant Cell Tumor of the Tendon Sheath (GCT-TS)
Brief Title: Tenosynovial Giant Cell Tumors (TGCT) Observational Platform Project
Acronym: TOP
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Optimapharm (Industry)
Responsible Party: Sponsor
Other Study IDs: DS-ONC-01-15-EU
Record Dates: First submitted 2016-10-24; First posted 2016-10-28 (Estimated); Results first posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-01

CONDITIONS: Giant Cell Tumors
Keywords: Tenosynovial Giant Cell Tumors; Disease registry; Routine clinical practice; Real World Evidence
MeSH Terms: conditions — Giant Cell Tumors; Synovitis, Pigmented Villonodular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
TGCT is a rare disease that is difficult to manage, surgical resection is the primary treatment currently available. To date no disease registry exists and there is little data available detailing the management of patients with diffuse TGCT (d-TGCT), the burden of d-TGCT for patients (including pain, joint stiffness, swelling, reduced mobility and quality of life) or the economic impact of d-TGCT.

This study aims to collect data by an observational disease registry involving no intervention to the patient or changes to investigators treatment decisions.

DETAILED DESCRIPTION:
GCT is a rare, benign, but potentially locally aggressive and recurrent disease. Treatment pattern and treatment initiation, continuation or changes are solely at the discretion of the physician and the patient.

There will be no attempt to influence the prescribing patterns of any individual treating physician. All medication will be prescribed in the usual standard of care and will not be provided by the study sponsor.

Participation in the study will in no way influence payment or reimbursement for any treatment received by patients during the study.

It is the responsibility of the investigator and his study staff to enter all relevant patient data required for this registry in the electronic Case Report Form (eCRF) and in the patients' medical records.

Approximately 15 sites from up to 6 European Countries (France, Germany, Italy, The Netherlands, Spain and United Kingdom) and 4 sites from the US are planned to participate. The sites will be specialized sites that treat d-TGCT regularly.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent for participation in the study (ICF)
* Patients with d-TGCT (diagnosed histologically) confirmed naïve or recurrent case

Exclusion Criteria:

* As this is a non interventional study, no explicit exclusion criteria have been defined

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study enrolled patients with d-TGCT.
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2016-11-18 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2021-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (15):
- United States (4):
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Medizinische Universität Graz, Graz, Austria
- CHU Nantes, Nantes, France
- Westdeutsches Tumorzentrum, Essen, Germany
- Italy (2):
  - Istituto Ortopedico Rizzoli, Bologna
  - Istituto Nazionale Tumori-Foundazione IRCCS, Milan
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - Radboud universitair medisch centrum, Nijmegen
- Spain (2):
  - Hospital Sant Pau, Barcelona
  - Hospital Universitario Virgen del Rocio, Seville
- United Kingdom (2):
  - The Royal Marsden Hospital, London
  - Nuffield Orthopaedic Centre, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palmerini E, Healey JH, Bernthal NM, Bauer S, Schreuder H, Leithner A, Martin-Broto J, Gouin F, Lopez-Bastida J, Gelderblom H, Staals EL, Mercier F, Laeis P, Ye X, van de Sande M. Tenosynovial Giant Cell Tumor Observational Platform Project (TOPP) Registry: A 2-Year Analysis of Patient-Reported Outcomes and Treatment Strategies. Oncologist. 2023 Jun 2;28(6):e425-e435. doi: 10.1093/oncolo/oyad011. PMID 36869793
- [Derived] Bernthal NM, Spierenburg G, Healey JH, Palmerini E, Bauer S; TOPP Study Group; Gelderblom H, Staals EL, Lopez-Bastida J, Fronk EM, Ye X, Laeis P, van de Sande MAJ. The diffuse-type tenosynovial giant cell tumor (dt-TGCT) patient journey: a prospective multicenter study. Orphanet J Rare Dis. 2021 Apr 29;16(1):191. doi: 10.1186/s13023-021-01820-6. PMID 33926503

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 183 participants who met all eligibility criteria were enrolled in the study at 12 sites in Europe and the United States.
Pre-assignment Details: All participants with diffuse TGCT (diagnosed histologically) with a confirmed primary diagnosis or recurrent case were enrolled.
Groups:
- Tenosynovial Giant Cell Tumors: All participants with diffuse tenosynovial giant cell tumors (d-TGCT) who were enrolled in the study.
Period: Overall Study
Arm/Group | Tenosynovial Giant Cell Tumors
Started (Baseline Analysis Set and All Documented Patient Set) | 183
Full Analysis Set | 176
Completed | 168
Not Completed | 15
Not completed — Lost to Follow-up | 8
Not completed — Death | 1
Not completed — Withdrawal by Subject | 4
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Population: Demographic and baseline characteristics were assessed in the Full Analysis Set.
Arm/Group | Tenosynovial Giant Cell Tumors
Number analyzed (Participants) | 176
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.5 (14.3)
Age, Customized [Count of Participants; unit: Participants]
  <40 years | 78
  ≥40 and <60 years | 69
  ≥60 years | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108
  Male | 68
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Austria | 10
  Netherlands | 61
  United States | 34
  Italy | 38
  United Kingdom | 3
  France | 4
  Germany | 12
  Spain | 14
Tumor location/affected joint [Count of Participants; unit: Participants]
  Knee joint | 120
  Ankle joint | 18
  Hip | 12
  Shoulder joint | 8
  Foot | 7
  Elbow joint | 4
  Wrist joint | 3
  Hand | 3
  Temporomandibular | 1
Current symptoms [Count of Participants; unit: Participants]
  Pain | 138
  Limited range of movement | 116
  Swelling | 111
  Stiffness | 99
  Patient unable to judge | 0
Most disturbing symptom [Count of Participants; unit: Participants]
  Pain | 86
  Stiffness | 13
  Swelling | 18
  Limited range of movement | 32
  Patient unable to judge | 16
  Not applicable | 8
  Missing | 3
Number of participants with current symptoms [Count of Participants; unit: Participants]
  4 current symptoms | 60
  3 current symptoms | 36
  2 current symptoms | 47
  Unknown/missing | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants According to the Management Plan in Patients With Diffuse TGCT (d-TGCT)
Description: The management plan received among the patients was collected from information routinely recorded in the patient files / medical records.
Time Frame: Baseline up to end of observation period (approximately 2 years)
Population: Management plans were assessed in participants with available data in the Full Analysis Set. Participants may have be included in more than one category.
Measure: Count of Participants; unit: Participants
Groups:
- Baseline: All participants with diffuse tenosynovial giant cell tumors (d-TGCT) who were enrolled at baseline in the study.
- Within 1st Year: Participants with diffuse tenosynovial giant cell tumors (d-TGCT) who were assessed within 1st year of the study.
- Within 2nd Year: Participants with diffuse tenosynovial giant cell tumors (d-TGCT) who were assessed within 2nd year of the study.
Arm/Group | Baseline | Within 1st Year | Within 2nd Year
Number analyzed (Participants) | 176 | 173 | 173
Participants
  Any prior or concomitant therapies for managing TGCT-related symptoms | 94 | NA — This parameter was only assessed at Baseline. | NA — This parameter was only assessed at Baseline.
  Any changes to concomitant therapies for managing TGCT-related symptoms since the last visit | NA — This parameter was based on changes since last visit and was only assessed within the 1st year and within the 2nd year. | 43 | 19
  Any changes to TGCT treatment (including also planned treatments) since the last visit | NA — This parameter was based on changes since last visit and was only assessed within the 1st year and within the 2nd year. | 74 | 61

2. Primary Outcome: Number of Participants According to the Current TGCT Treatment Plan in Patients With Diffuse TGCT (d-TGCT)
Description: The current TGCT treatment plan among the patients was collected from information routinely recorded in the patient files / medical records.
Time Frame: Baseline up to end of observation period (approximately 2 years)
Population: The current treatment plan (currently being treated or planned) was assessed in participants with no changes at any data collection point where the data of the previous reported data collection point is being reported in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline | Within 1st Year | Within 2nd Year
Number analyzed (Participants) | 176 | 173 | 173
Participants
  Wait and see | 79 | 77 | 105
  Currently being treated or planned to be treated | 97 | 85 | 65
  Unknown/Missing | 0 | 11 | 3

3. Primary Outcome: Number of Participants Based on Type of Treatment Plan in Patients With Diffuse TGCT (d-TGCT)
Description: Type of treatment plan received among the patients was collected from information routinely recorded in the patient files / medical records.
Time Frame: Baseline up to end of observation period (approximately 2 years)
Population: Type of treatment plans were assessed in participants with available data in the Full Analysis Set. Participants may have be included in more than one category.
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline | Within 1st Year | Within 2nd Year
Number analyzed (Participants) | 176 | 173 | 173
Participants
  Radiotherapy | 5 | 1 | 0
  90Yttrium therapy | 1 | 1 | 0
  Systemic therapy | 48 | 16 | 8
  Surgery | 42 | 40 | 25
  Future surgery required | 5 | 2 | 0
  No current or planned treatment | 79 | 77 | 105
  Unchanged therapy | 0 | 36 | 35

4. Primary Outcome: Number of Participants Based on Status of Treatment Plan in Patients With Diffuse TGCT (d-TGCT)
Description: The status of treatment plan among the patients was collected from information routinely recorded in the patient files / medical records.
Time Frame: Baseline up to end of observation period (approximately 2 years)
Population: Status of treatment plan was assessed in participants currently being treated or planned to be treated in the Full Analysis Set. Participants with different reported treatment plans during the period (e.g. participants who may have switched treatment plans) are counted as 'currently being treated or planned to be treated' in the corresponding period.
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline | Within 1st Year | Within 2nd Year
Number analyzed (Participants) | 99 | 61 | 32
Participants
  Planned | 50 | 9 | 9
  Current | 44 | 50 | 23
  Missing | 5 | 2 | 0

5. Primary Outcome: Number of Participants Based on Type of Current TGCT Treatment in Patients With Diffuse TGCT (d-TGCT)
Description: Type of current TGCT treatment among the patients was collected from information routinely recorded in the patient files / medical records.
Time Frame: Baseline up to end of observation period (approximately 2 years)
Population: Status of treatment plan was assessed in participants currently being treated in the Full Analysis Set. Participants may have been included in more than one category.
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline | Within 1st Year | Within 2nd Year
Number analyzed (Participants) | 44 | 50 | 23
Participants
  90Yttrium therapy | 0 | 1 | 0
  Systemic therapy | 37 | 12 | 8
  Surgery | 7 | 37 | 17

6. Primary Outcome: Number of Participants Based on Tumor Severity Classification at Baseline Based on MRI in Patients With Diffuse TGCT (d-TGCT)
Description: Tumor severity classification was collected from information routinely recorded in the patient files / medical records. ). Tumor severity classification was based on MRI. In this classification scheme, moderate diffuse TGCT is characterized by intra- and/or extra-articular disease, without or with involvement of muscle/tendinous tissue/ligaments. Severe diffuse TGCT is characterized by intra- and extra-articular involvement and involvement of at least one of the 3 structures (muscle/tendinous tissue/ligaments).
Time Frame: at Baseline
Population: Tumor severity was assessed in participants in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Tenosynovial Giant Cell Tumors
Number analyzed (Participants) | 176
Participants
  Moderate diffuse | 66
  Severe diffuse | 90
  Not assessable | 20

7. Primary Outcome: Number of Cases With Complications Due to Surgery in Patients With Diffuse TGCT (d-TGCT)
Description: Complications due to surgery were collected from information routinely recorded in the patient files / medical records.
Time Frame: at Baseline (prior to any d-TGCT therapy)
Population: Complications were assessed among participants with documented surgeries.
Measure: Number; unit: surgical cases
Units Other Than Participants: Surgeries
Arm/Group | Tenosynovial Giant Cell Tumors
Number analyzed (Participants) | 134
Number analyzed (Surgeries) | 210
surgical cases | 9

8. Primary Outcome: Number of Participants With Tumor Recurrence at Baseline in Patients With Diffuse TGCT (d-TGCT)
Description: Tumor recurrence was collected from information routinely recorded in the patient files / medical records.
Time Frame: at Baseline
Population: Tumor recurrence was assessed in participants with available baseline data in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Groups:
- Participants With Tumor Recurrence: All participants with diffuse tenosynovial giant cell tumors (d-TGCT) with tumor recurrence.
Arm/Group | Participants With Tumor Recurrence
Number analyzed (Participants) | 78
Participants
  1 recurrence | 40
  2 recurrences | 18
  3 recurrences and more | 19
  Missing | 1

9. Primary Outcome: Time Since Most Recent Tumor Recurrence Until Baseline in Patients With Diffuse TGCT (d-TGCT)
Description: Time since most recent tumor recurrence was collected from information routinely recorded in the patient files / medical records.
Time Frame: at Baseline
Population: Time since last recent tumor recurrence until baseline was assessed in participants with available baseline data in the Full Analysis Set.
Measure: Median (Full Range); unit: months
Groups:
- Tenosynovial Giant Cell Tumors: All participants with diffuse tenosynovial giant cell tumors (TGCT) who were enrolled in the study.
Arm/Group | Tenosynovial Giant Cell Tumors
Number analyzed (Participants) | 77
months | 12.55 [0.03 to 137.49]

10. Primary Outcome: Time From Baseline to First Tumor Recurrence in Patients With Diffuse TGCT (d-TGCT)
Description: Time from baseline to first tumor recurrence was collected from information routinely recorded in the patient files / medical records.
Time Frame: Baseline up to end of observation period (approximately 2 years)
Population: Time from baseline to first tumor recurrence was assessed in participants with available data in the Full Analysis Set.
Measure: Median (Full Range); unit: months
Groups:
- Within 1st Year: Participants with diffuse tenosynovial giant cell tumors (d-TGCT) who were assessed for tumor recurrence within 1st year of the study.
- Within 2nd Year: Participants with diffuse tenosynovial giant cell tumors (d-TGCT) who were assessed for tumor recurrence within 2nd year of the study.
- Tenosynovial Giant Cell Tumors: All participants with diffuse tenosynovial giant cell tumors (d-TGCT) who were assessed for tumor recurrence within the whole observation period.
Arm/Group | Within 1st Year | Within 2nd Year | Tenosynovial Giant Cell Tumors
Number analyzed (Participants) | 6 | 9 | 15
months | 8.4 [2 to 15] | 19.0 [12 to 24] | 14.8 [2 to 24]

11. Primary Outcome: Mean Brief Pain Inventory (BPI) Pain Severity and Interference Score From Baseline Through 24 Months
Description: The BPI short form is a self administered questionnaire that assesses severity of pain, impact of pain on daily function, location of pain, pain medications and amount of pain relief in the past 24 hours or the past week. The BPI pain severity and interference score ranges from 0 (pain does not interfere) to 10 (pain completely interferes), where lower scores indicate better clinical outcome.
Time Frame: Baseline up to end of observation period (approximately 2 years)
Population: Brief Pain Inventory Pain Severity and Pain Interference were assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline: Participants with diffuse tenosynovial giant cell tumors (d-TGCT) who had BPI Pain Severity and Pain Interference assessments conducted at baseline.
- 6 Months: Participants with diffuse tenosynovial giant cell tumors (d-TGCT) who had BPI Pain Severity and Pain Interference assessments conducted at 6 months.
- 12 Months: Participants with diffuse tenosynovial giant cell tumors (d-TGCT) who had BPI Pain Severity and Pain Interference assessments conducted at 12 months.
- 18 Months: Participants with diffuse tenosynovial giant cell tumors (d-TGCT) who had BPI Pain Severity and Pain Interference assessments conducted at 18 months.
- 24 Months: Participants with diffuse tenosynovial giant cell tumors (d-TGCT) who had BPI Pain Severity and Pain Interference assessments conducted at 24 months.
Arm/Group | Baseline | 6 Months | 12 Months | 18 Months | 24 Months
Number analyzed (Participants) | 166 | 130 | 125 | 125 | 132
score on a scale
  Brief Pain Inventory Pain Severity | 3.35 (2.36) | 3.12 (2.26) | 3.15 (2.22) | 3.05 (2.30) | 2.60 (2.19)
  Brief Pain Inventory Pain Interference: number analyzed (Participants) | 165 | 129 | 123 | 122 | 132
  Brief Pain Inventory Pain Interference | 2.97 (2.65) | 2.94 (2.56) | 2.80 (2.44) | 2.80 (2.47) | 2.53 (2.57)

12. Primary Outcome: Mean Worst Stiffness Score From Baseline Through 24 Months
Description: The Worst Stiffness numerical rating scale (NRS) is a one-item self-administered, patient-reported outcome questionnaire assessing the "worst" stiffness in the last 24 hours. The NRS for this item ranges from 0 ("no stiffness") to 10 ("stiffness as bad as you can imagine"), where lower scores indicate better clinical outcome.
Time Frame: Baseline up to end of observation period (approximately 2 years)
Population: Worst stiffness was assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline: Participants with diffuse tenosynovial giant cell tumors (d-TGCT) who assessed worst stiffness in last 24 hours (patient reported outcome) at baseline.
- 6 Months: Participants with diffuse tenosynovial giant cell tumors (d-TGCT) who assessed worst stiffness in last 24 hours (patient reported outcome) at 6 months.
- 18 Months: Participants with diffuse tenosynovial giant cell tumors (d-TGCT) who assessed worst stiffness in last 24 hours (patient reported outcome) at 18 months.
- 24 Months: Participants with diffuse tenosynovial giant cell tumors (d-TGCT) who assessed worst stiffness in last 24 hours (patient reported outcome) at 24 months.
Arm/Group | Baseline | 6 Months | 12 Months | 18 Months | 24 Months
Number analyzed (Participants) | 164 | 132 | 129 | 125 | 133
score on a scale | 4.4 (2.8) | 4.2 (2.6) | 4.2 (2.8) | 4.2 (2.7) | 3.9 (2.7)

13. Primary Outcome: Mean PROMIS Physical Function Score From Baseline Through 24 Months
Description: PROMIS® (Patient-Reported Outcomes Measurement Information System) is a set of person-centered measures that evaluates and monitors physical, mental, and social health. Physical function scores range from 0 (worst physical function) to 100 (best physical function, where higher scores indicate better clinical outcome.
Time Frame: Baseline up to end of observation period (approximately 2 years)
Population: PROMIS physical function was assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline: Participants with diffuse tenosynovial giant cell tumors (d-TGCT) who assessed their physical function at baseline.
- 6 Months: Participants with diffuse tenosynovial giant cell tumors (d-TGCT) who assessed their physical function at 6 months.
- 12 Months: Participants with diffuse tenosynovial giant cell tumors (d-TGCT) who assessed their physical function at 12 months.
- 18 Months: Participants with diffuse tenosynovial giant cell tumors (d-TGCT) who assessed their physical function at 18 months.
- 24 Months: Participants with diffuse tenosynovial giant cell tumors (d-TGCT) who assessed their physical function at 24 months.
Arm/Group | Baseline | 6 Months | 12 Months | 18 Months | 24 Months
Number analyzed (Participants) | 168 | 132 | 130 | 126 | 136
score on a scale | 41.9 (8.2) | 41.6 (9.2) | 43.2 (9.3) | 42.2 (8.8) | 43.0 (9.0)

14. Secondary Outcome: Mean EuroQol Questionnaire (EQ) of 5 Dimensions (5D) Index Score and EQ Visual Analog Scale Score From Baseline Through 24 Months
Description: The EQ-5D-5L questionnaire measures the patient's quality of life (QoL) based on the 5 dimensions mobility, self care, usual activities, pain/discomfort, and anxiety/depression. The EQ-5D index score ranges from 0 (worst QoL) to 1 (best QoL), where lower scores indicate worse clinical outcome. The EQ-5D VAS reports patient's self rated health ranging from 0 (worst health) to 100 (best health you can imagine), where lower scores indicate worse clinical outcome.
Time Frame: Baseline up to end of observation period (approximately 2 years)
Population: Quality of life assessed by EQ-5D index score was assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Baseline: Participants with diffuse tenosynovial giant cell tumors (d-TGCT) who assessed their quality of life at baseline.
- 6 Months: Participants with diffuse tenosynovial giant cell tumors (d-TGCT) who assessed their quality of life at 6 months.
- 12 Months: Participants with diffuse tenosynovial giant cell tumors (d-TGCT) who assessed their quality of life at 12 months.
- 18 Months: Participants with diffuse tenosynovial giant cell tumors (d-TGCT) who assessed their quality of life at 18 months.
- 24 Months: Participants with diffuse tenosynovial giant cell tumors (d-TGCT) who assessed their quality of life at 24 months.
Arm/Group | Baseline | 6 Months | 12 Months | 18 Months | 24 Months
Number analyzed (Participants) | 168 | 133 | 130 | 126 | 135
score on a scale
  EQ-5D Index Score: number analyzed (Participants) | 166 | 132 | 128 | 126 | 133
  EQ-5D Index Score | 0.714 (0.20) | 0.742 (0.18) | 0.740 (0.20) | 0.741 (0.20) | 0.746 (0.21)
  EQ-5D VAS: number analyzed (Participants) | 168 | 133 | 130 | 125 | 135
  EQ-5D VAS | 69.3 (20.95) | 69.0 (19.84) | 73.0 (18.23) | 69.8 (20.53) | 71.7 (20.74)

15. Secondary Outcome: Mean Number of General Practitioner, Specialist, or Physical Therapy Visits to Assess the Health Resource Utilization in Patients With Diffuse TGCT Through 24 Months
Description: Health resource utilization was assessed by mean number of general practitioner visits, specialist visits, and physical therapy sessions. In addition, the mean number of days in rehabilitation and the number of work days missed were also reported.
Time Frame: 13-24 months before baseline up to end of observation period (approximately 2 years)
Population: Health resource utilization was assessed in participants with available data in the Full Analysis Set.
Measure: Mean (Standard Deviation); unit: visits
Groups:
- 13-24 Months Before Baseline: Participants with diffuse tenosynovial giant cell tumors (d-TGCT) who were assessed and categorized by tumor status within 13-24 months before baseline.
- 1-12 Months Before Baseline: Participants with diffuse tenosynovial giant cell tumors (d-TGCT) who were assessed and categorized by tumor status within 1-12 months before baseline.
- Within 1st Year: Participants with diffuse tenosynovial giant cell tumors (d-TGCT) who were assessed and categorized by tumor status within 1st year of the study.
- Within 2nd Year: Participants with diffuse tenosynovial giant cell tumors (d-TGCT) who were assessed and categorized by tumor status within 2nd year of the study.
- Within Whole 2-year Period: All participants with diffuse tenosynovial giant cell tumors (d-TGCT) who were assessed and categorized by tumor status within the whole observation period.
Arm/Group | 13-24 Months Before Baseline | 1-12 Months Before Baseline | Within 1st Year | Within 2nd Year | Within Whole 2-year Period
Number analyzed (Participants) | 176 | 176 | 176 | 173 | 176
visits
  General practitioner visits | 3.9 (4.80) | 3.0 (4.60) | 3.8 (4.03) | 3.3 (4.83) | 4.7 (5.71)
  Specialists visits | 7.0 (8.55) | 5.2 (5.89) | 4.1 (3.76) | 2.6 (2.80) | 5.1 (4.82)
  Physical therapy sessions | 20.3 (22.93) | 25.4 (27.96) | 17.7 (14.34) | 33.1 (31.12) | 31.3 (32.44)

16. Secondary Outcome: Median Number of Days in Rehabilitation and Work Days Missed in Patients With Diffuse TGCT Through 24 Months
Description: The median number of days in rehabilitation and the number of work days missed were also reported.
Time Frame: 13-24 months before baseline up to end of observation period (approximately 2 years)
Population: Number of days in rehabilitation was assessed in the Full Analysis Set. A participant could have documented days in rehabilitation for the 1st year visit as well as for the 2nd year visit which resulted in a sum greater than the single results per visit/year.
Measure: Median (Full Range); unit: days
Arm/Group | 13-24 Months Before Baseline | 1-12 Months Before Baseline | Within 1st Year | Within 2nd Year | Within Whole 2-year Period
Number analyzed (Participants) | 176 | 176 | 176 | 173 | 176
days
  Days in rehabilitation | 15 [3 to 60] | 15 [1 to 60] | 12 [1 to 45] | 20 [4 to 150] | 16 [1 to 151]
  Work days missed | 25.50 [0.5 to 180] | 16 [1 to 180] | 6 [1 to 180] | 8 [1 to 73] | 10 [1 to 180]

17. Secondary Outcome: Overall TGCT Outcome Status in Patients With Diffuse TGCT (d-TGCT)
Description: TGCT outcome status was collected from information routinely recorded in the patient files / medical records.
Time Frame: At end of observation period (approximately 2 years post-baseline)
Population: TGCT outcome status was assessed in participants with available data in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Tenosynovial Giant Cell Tumors
Number analyzed (Participants) | 166
Participants
  TCGT status at end of observational period: No evidence of disease (NED) | 39
  TCGT status at end of observational period: Radiological residual disease | 107
  TCGT status at end of observational period: Radiological recurrent disease | 20
  TCGT status at end of observational period: Missing | 10
  NED (only pts with NED): With complaints: number analyzed (Participants) | 39
  NED (only pts with NED): With complaints | 21
  NED (only pts with NED): Without complaints: number analyzed (Participants) | 39
  NED (only pts with NED): Without complaints | 18
  NED (only pts with NED): Missing: number analyzed (Participants) | 39
  NED (only pts with NED): Missing | 0
  Radiological residual disease (only pts with radiological residual disease): Watchful waiting: number analyzed (Participants) | 106
  Radiological residual disease (only pts with radiological residual disease): Watchful waiting | 84
  Radiological residual disease (only pts with radiological residual disease): Awaiting surgery: number analyzed (Participants) | 106
  Radiological residual disease (only pts with radiological residual disease): Awaiting surgery | 4
  Radiological residual disease (only pts with radiological residual disease): Awaiting medication: number analyzed (Participants) | 106
  Radiological residual disease (only pts with radiological residual disease): Awaiting medication | 16
  Radiological residual disease (only pts with radiological residual disease):Awaiting other treatment: number analyzed (Participants) | 106
  Radiological residual disease (only pts with radiological residual disease):Awaiting other treatment | 2
  Radiological residual disease (only pts with radiological residual disease): Missing: number analyzed (Participants) | 106
  Radiological residual disease (only pts with radiological residual disease): Missing | 1
  Radiological recurrent disease (only pts with radiological recurrent disease): Watchful waiting: number analyzed (Participants) | 20
  Radiological recurrent disease (only pts with radiological recurrent disease): Watchful waiting | 12
  Radiological recurrent disease (only pts with radiological recurrent disease): Awaiting surgery: number analyzed (Participants) | 20
  Radiological recurrent disease (only pts with radiological recurrent disease): Awaiting surgery | 6
  Radiological recurrent disease (only pts with radiological recurrent disease): Awaiting medication: number analyzed (Participants) | 20
  Radiological recurrent disease (only pts with radiological recurrent disease): Awaiting medication | 1
  Radiological recurrent disease (only pts with radiological recurrent): Awaiting other treatment: number analyzed (Participants) | 20
  Radiological recurrent disease (only pts with radiological recurrent): Awaiting other treatment | 1
  Radiological recurrent disease (only pts with radiological recurrent disease): Missing: number analyzed (Participants) | 20
  Radiological recurrent disease (only pts with radiological recurrent disease): Missing | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were not assessed in this non-interventional study.
Description: Treatment-emergent adverse events and serious adverse events were not assessed in this non-interventional study. Adverse drug reactions suspected to be related to pexidartinib were only collated for patients from the United States.
Groups:
- Overall: All participants with diffuse tenosynovial giant cell tumors (d-TGCT) who were enrolled in the study.
Arm/Group | Overall
All-Cause Mortality (participants affected / at risk) | 1/183
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
This was an observational study and the quality of data has not been verified 100%. Baseline data were checked during on-site visits for all patients enrolled in Europe. Due to the COVID-19 pandemic, the planned on-site monitoring visits in the US could not be performed. Instead, more frequent and detailed remote visits were performed for these sites. Follow-up data for all patients were regularly monitored remotely. A certain amount of incorrect/incomplete data has to be assumed for all sites.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-15): https://cdn.clinicaltrials.gov/large-docs/88/NCT02948088/Prot_SAP_000.pdf